CLINICAL TRIAL: NCT01954654
Title: Effectiveness of Accelerated Intervention With Custom-made Compression Sleeve in Women With Mild and Moderate Arm Lymphedema Secondary to Breast Cancer Treatment
Brief Title: Effectiveness of Accelerated Intervention With Compression Sleeve in Mild and Moderate Breast Cancer-related Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mette Brodersen Jerver (Other)
Responsible Party: Sponsor-Investigator, Mette Brodersen Jerver, Physiotherapist, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-58-0010
Record Dates: First submitted 2013-09-29; First posted 2013-10-07 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Accelerated treatment (Experimental)
  Interventions: Device: Custom-made compression sleeve and -gauntlet; Other: Educational information, recommendation and instruction
- Standard treatment (Active Comparator)
  Interventions: Device: Custom-made compression sleeve and -gauntlet; Other: Educational information, recommendation and instruction

INTERVENTIONS:
Device: Custom-made compression sleeve and -gauntlet — Device: Compression garments worn for a minimum of six hours per day
  Other Names: Jobst Elvarex
Other: Educational information, recommendation and instruction — Educational information and recommendations about lymphedema and skin care. Instruction in physical exercises to enhance the lymph flow

SUMMARY:
The purpose of this study is to determine whether accelerated treatment with custom-made compression sleeve is more effective than standard procedure in the treatment of mild and moderate arm lymphedema secondary to primary cancer treatment.

DETAILED DESCRIPTION:
Use of a custom-made compression sleeve is an initial treatment of mild and moderate arm lymphedema secondary to primary breast cancer treatment. The compression sleeve improves the flow of lymph fluid out of the arm, reduces the swelling, and prevents progression of the lymphedema in the future.

Early intervention is recommended though early is not well-defined in literature. The purpose of this study is to evaluate reduction of excess limb volume and changes in arm disability and clinical symptoms in accelerated treatment with compression sleeve compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be refered for the first time due to unilateral arm lymphedema secondary to primary unilateral breast cancer treatment
* Participants must be ≥ 2 months after chemo- and radiotherapy
* Participants must have ELV ≥10% and < 30% and/or > 2 cm difference between the circumference of the two arms at minimum one circumference due to lymphedema
* Participants must be motivated for treatment with compression sleeve and -gauntlet
* Participants live in and around Aarhus, Denmark

Exclusion Criteria:

* Known metastatic disease
* Contraindication for treatment with compression sleeve
* Upper extremity deep venous thrombosis
* Previously use of compression sleeve
* Known contact allergy to latex
* Unable to fill in questionnaire and/or comply with treatment due to lacking Danish language skills, mental state or psychological condition

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Change of excess limb volume (ELV) | 8 weeks follow-up
  ELV in the affected arm compared to the non-affected arm. ELV described as both absolute volume in ml and relative volume in percent

SECONDARY OUTCOMES:
Changes in arm disability | 8 weeks follow-up
  Measured with Disabilities of Arm, Shoulder, and Hand (DASH)
Changes in subjective symptoms (pain, tension, and heaviness) | 8 weeks follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Fysioterapi- og Ergoterapisfdelingen, Aarhus, Aarhus, Denmark